CLINICAL TRIAL: NCT03405116
Title: Neonatal and Long Term Outcomes of Preterm Born Children in Flanders
Brief Title: Prediction Tool for Premature Labour and Neonatal Outcome
Acronym: PRETURN
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201732321 (BC-00466)
Record Dates: First submitted 2017-11-23; First posted 2018-01-19 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years

SUMMARY:
A register and prediction model will be developed to predict the outcome of preterm labour and birth.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 24 weeks 0 days and 33 weeks and 6 days, and their preterm born children

Exclusion Criteria:

* Patients who choose not to participate in the research.
* Intra-uterine prelabour fetal death.
* Fetuses or neonates with a major congenital disorder. Major is defined as a disorder that has an impact on neonatal respiratory and cerebral outcome and/or long-term outcome.
* Postpartum transfer/outborn.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women visiting the maternity ward suffering from symptoms of preterm birth.
Sampling Method: Probability Sample
Enrollment: 2037 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Register | 2017 - 2030
  A multicentre, multidisciplinary register will be created to provide a source of valuable information on obstetrical and neonatal practices and link them with obstetrical, neonatal and long-term outcomes of preterm labour and birth
Prediction model | 2017 - 2030
  The prediction tool for true preterm labour (TPL) will be developed using individual risk factors, symptomatology, tocography, cervical change and a biomarker test, followed by a decision-making model, both based on individual data, evidence and experience.

SECONDARY OUTCOMES:
The interval between starting corticosteroids and delivery | 2012-2020
  The interval between administration of antenatal corticosteroids and birth will be assessed and will be related to the short and long term outcome of preterm born children

CONTACTS AND LOCATIONS:
Overall Officials: Kristien Roelens, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital - Women's Clinic, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dehaene I, Scheire E, Steen J, De Coen K, Decruyenaere J, Smets K, Roelens K. Obstetrical characteristics and neonatal outcome according to aetiology of preterm birth: a cohort study. Arch Gynecol Obstet. 2020 Oct;302(4):861-871. doi: 10.1007/s00404-020-05673-5. Epub 2020 Jul 3. PMID 32621250